CLINICAL TRIAL: NCT05022251
Title: Identifying Pain Generators and Potentiators of Residual Complaints Following Lumbar Discectomy
Acronym: DISC-PAIN
Status: Terminated | Type: Observational
Why Stopped: Diffculty recruiting patients, limited timeframe to complete project
Sponsor: University Ghent (Other)
Collaborators: Research Foundation Flanders (Other)
Responsible Party: Sponsor
Other Study IDs: BC-08041; 3F014119 (Other Grant/Funding Number: Research Foundation - Flanders (FWO))
Record Dates: First submitted 2021-05-12; First posted 2021-08-26 (Actual); Last update posted 2023-12-20 (Actual); Status verified 2023-12

CONDITIONS: Lumbar Radiculopathy; Central Sensitisation
Keywords: lumbar radiculopathy; discectomy; central sensitization
MeSH Terms: conditions — Radiculopathy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Lumbar radiculopathy: Lumbar radiculopathy patients (n=122), classified as ASA I to II without any symptoms of spinal cord compression (i.e. bilateral leg pain), who are scheduled for a first-time, single-level, unilateral lumbar discectomy.
  Interventions: Procedure: Lumbar discectomy
- Healthy controls: Sex, age, and BMI-matched healthy, pain-free control subjects (n=122) will be recruited for study participation.

INTERVENTIONS:
Procedure: Lumbar discectomy — surgically removing a hernia
  Groups: Lumbar radiculopathy

SUMMARY:
Lumbar discectomy (i.e. surgically removing a hernia) is frequently performed in Belgium to treat lumbar radiculopathy. Every year >12,000 interventions are performed with variable long-term results. The treatment success of this procedure varies and up to 41% of the patients report post-operative persistent pain complaints, and consequently suffer from failed back surgery syndrome (FBSS). Chronic complaints in FBSS following lumbar discectomy are usually treated with symptomatic interventions (including painkillers, neuromodulation, etc), rather than from a biopsychosocial perspective.

In order to develop a focused and effective treatment strategy, it is crucial to first gain insight into how persons with persistent complaints after lumbar discectomy differ from those without persistent symptoms. Different known contributing factors entail type of surgery, muscle and psychosocial impairments. Although in scientific and clinical literature it is assumed that dysfunctional pain processing also plays an important mechanistic role in FBSS, there is a lack of research to support this. However, this knowledge is crucial to depict the full mechanistic picture of pain generators and potentiators in FBSS.

Therefore, we will examine whether residual complaints persisting following lumbar discectomy can be accounted for by underlying dysfunctional pain processing and whether a clinical classification algorithm can be used to identify the predominant pain mechanism in these patients.

ELIGIBILITY:
Inclusion Criteria:

* Dutch speaking
* Body mass index below 35kg/m²
* Lumbar radiculopathy patients, classified as ASA I to II without any symptoms of spinal cord compression (i.e. bilateral leg pain), who are scheduled for a first-time, single-level, unilateral lumbar discectomy
* Healthy, pain-free controls (score 0 on a visual analogue scale from 0 to 100)

Exclusion Criteria:

* Female participants will be excluded if pregnant, lactating or <1 year postnatal
* Having (a history) of severe medical disorders either respiratory (e.g. cystic fibrosis), orthopedic (e.g. whiplash trauma), neurologic (e.g. cerebrovascular incident), cardiovascular (e.g. severe hypertension), endocrinological (e.g. diabetes), psychiatric (e.g. post-traumatic stress disorder
* Having a history of spinal surgery (e.g. discectomy), spinal traumata (e.g. vertebral fracture) or severe spinal deformities (e.g. spondylolisthesis)
* Having a pacemaker or defibrillator
* Healthy controls will be excluded if having suffered low back pain in the preceding year of score 2 or higher on the visual analog scale and which limited their activities of daily living or for which they consulted a (para)medic.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Lumbar radiculopathy patients scheduled for first-time, single level, unilateral lumbar discectomy.
  Sex, age, and BMI matched healthy controls.
Sampling Method: Non-Probability Sample
Enrollment: 1 (Actual)
Dates: Start 2021-10-01 (Actual); Primary Completion 2023-10-31 (Actual); Study Completion 2023-10-31 (Actual)

PRIMARY OUTCOMES:
Quantitative sensory testing (QST) - electrical detection threshold | Change from baseline (T1) at 3 months after surgery (T2)
  Determination of sensory detection thresholds in response to electrical stimuli which are delivered transcutaneously over the n. suralis and n. medianus, recorded in mA.
Quantitative sensory testing (QST) - electrical pain threshold | Change from baseline (T1) at 3 months after surgery (T2)
  Determination of sensory pain threshold in response to electrical stimuli which are delivered transcutaneously over the n. suralis and n. medianus, recorded in mA.
Quantitative sensory testing (QST) - thermal detection threshold | Change from baseline (T1) at 3 months after surgery (T2)
  Determination of sensory detection thresholds in response to thermal stimuli which are delivered to the skin using a thermode, recorded in °C:
  * cold detection threshold
  * warmth detection threshold
Quantitative sensory testing (QST) - thermal pain threshold | Change from baseline (T1) at 3 months after surgery (T2)
  Determination of sensory pain thresholds in response to thermal stimuli which are delivered to the skin using a thermode, recorded in °C:
  * cold pain threshold
  * heat pain threshold
Quantitative sensory testing (QST) - discrimination between thermal stimuli | Change from baseline (T1) at 3 months after surgery (T2)
  Determination of the number of paradoxical heat sensations in response to alternating cold and warm stimuli delivered to the skin using a thermode.
Quantitative sensory testing (QST) - tactile detection threshold | Change from baseline (T1) at 3 months after surgery (T2)
  Determination of tactile detection threshold, assessed using Von Frey monofilaments, recorded in mN
Quantitative sensory testing (QST) - mechanical pain threshold | Change from baseline (T1) at 3 months after surgery (T2)
  Determination of mechanical pain threshold, assessed using pinprick stimulators, recorded in mN
Quantitative sensory testing (QST) - sensitivity to pressure stimuli | Change from baseline (T1) at 3 months after surgery (T2)
  Determination of pressure pain threshold, assessed using pressure algometry, recorded in kg
Quantitative sensory testing (QST) - temporal summation of electrical stimuli | Change from baseline (T1) and 3 months after surgery (T2)
  Determination of temporal summation in response to electrical stimuli delivered transcutaneously over the skin of the n. suralis and n. medianus.
  The numerical pain rating in response to these stimuli (range 0 - 100) will be recorded.
Quantitative sensory testing (QST) - temporal summation of mechanical stimuli | Change from baseline (T1) and 3 months after surgery (T2)
  Determination of temporal summation in response to mechanical stimuli delivered using a 256mN pinprick stimulator.
  The numerical pain rating in response to these stimuli (range 0 - 100) will be recorded.
Quantitative sensory testing (QST) - spinal hyperexcitability | Change from baseline (T1) and 3 months after surgery (T2)
  Determination of spinal hyperexcitability using the nociceptive flexion reflex (NFR; sensitization of spinal cord neurons), recorded in mA
Quantitative sensory testing (QST) - temporal summation of spinal hyperexcitability | Change from baseline (T1) and 3 months after surgery (T2)
  Determination of temporal summation of the nociceptive flexion reflex (NFR; sensitization of spinal cord neurons), recorded using a numeric pain rating scale (range 0 - 100)
Quantitative sensory testing - conditioned pain modulation | Change from baseline (T1) and 3 months after surgery (T2)
  Determination of condition pain modulation (aka. pain inhibits pain) by means of a heterotopic noxious counterstimulation paradigm. Test stimuli comprise of pressure pain threshold assessments and application of a heat stimulus (using a thermode) corresponding to a temperature eliciting a visual analog scale rating of 5/10. Test stimuli will be applied before, during and after the conditioning stimulus which is the immersion of the hand in a hot circulating water bath of 45.5°C.

SECONDARY OUTCOMES:
Central sensitization inventory | Baseline (T1)
  Self-report measure of signs and symptoms associated with central sensitization
Central sensitization inventory | 3 months after surgery (T2)
  Self-report measure of signs and symptoms associated with central sensitization
Douleur Neuropathique 4 Questionnaire | Baseline (T1)
  Clinician administered questionnaire for evaluation of signs and symptoms associated with neuropathic pain
Douleur Neuropathique 4 Questionnaire | 3 months after surgery (T2)
  Clinician administered questionnaire for evaluation of signs and symptoms associated with neuropathic pain
Pain catastrophizing scale | Baseline (T1)
  Self-report measure of pain perceptions and cognitions
Pain catastrophizing scale | 3 months after surgery (T2)
  Self-report measure of pain perceptions and cognitions
Pain vigilance and awareness questionnaire | Baseline (T1)
  Self-report measure assessing preoccupation with and attention to pain
Pain vigilance and awareness questionnaire | 3 months after surgery (T2)
  Self-report measure assessing preoccupation with and attention to pain
Oswestry disability index | Baseline (T1)
  Self-report measure evaluating low back pain related disability
Oswestry disability index | 3 months after surgery (T2)
  Self-report measure evaluating low back pain related disability
Tampa scale for kinesiophobia | Baseline (T1)
  Self-report measure assessing fear of movement
Tampa scale for kinesiophobia | 3 months after surgery (T2)
  Self-report measure assessing fear of movement
International physical activity questionnaire | Baseline (T1)
  Self-report measure of physical activity in preceeding 7 days
International physical activity questionnaire | 3 months after surgery (T2)
  Self-report measure of physical activity in preceeding 7 days
Patient-reported outcomes measurement information system | Baseline (T1)
  Self-report measure of health-related domains including:
  * physical functioning
  * anxiety
  * depression
  * fatigue
  * sleep disruption
  * participation in social activities
  * pain interference
Patient-reported outcomes measurement information system | 3 months after surgery (T2)
  Self-report measure of health-related domains including:
  * physical functioning
  * anxiety
  * depression
  * fatigue
  * sleep disruption
  * participation in social activities
  * pain interference
Brief Illness Perception Questionnaire | Baseline (T1)
  Self-report measure evaluating illness perceptions
Brief Illness Perception Questionnaire | 3 months after surgery (T2)
  Self-report measure evaluating illness perceptions
Pain Coping Inventory | Baseline (T1)
  Self-report measure assessing pain coping strategies
Pain Coping Inventory | 3 months after surgery (T2)
  Self-report measure assessing pain coping strategies

CONTACTS AND LOCATIONS:
Overall Officials: Jessica Van Oosterwijck, PhD, Study Director — Ghent University; Research Foundation Flanders
Locations (1):
- Ghent University (Hospital), Ghent, Belgium

IPD SHARING:
Plan to Share IPD: Undecided